CLINICAL TRIAL: NCT04773847
Title: The Clinical and Radiographic Outcomes of a 3D-printed Patient-specific Biomimetic Bone Substitute in Maxillofacial Indications: an Interventional, Multi-centred, Open-label, Post-market Clinical Investigation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mimetis Biomaterials S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/743
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Bone Regeneration

STUDY DESIGN:
Intervention Model Description: Since the studied medical device is a custom-made product, only one group is considered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MimetikOss 3D (Experimental)
  Interventions: Procedure: Surgical reconstruction of maxillofacial osseous defect with MimetikOss 3D.

INTERVENTIONS:
Procedure: Surgical reconstruction of maxillofacial osseous defect with MimetikOss 3D. — Surgical reconstruction of maxillofacial osseous defect with MimetikOss 3D.

SUMMARY:
The purpose of the study is to evaluate the clinical and radiographic outcome of MimetikOss 3D as a patient-specific bone substitute in regeneration of osseous defects in several maxillofacial indications. The primary objective is to evaluate the capacity of MimetikOss 3D to perform bone substitute requirements, i.e long-term regeneration of bony tissue in complex defects without detrimental resorption. The secondary main objectives are to assess the versatility of MimetikOss 3D by the variety of maxillofacial sites regenerated and the surgical technique improvement (in terms of surgery duration, blood loss, ease-of-use of the product and surgeon satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 years or over at the time of inclusion into the study;
* Ability to obtain written informed consent from the recipient;
* Patients in need of craniomaxillofacial bone regeneration;
* Ability and capacity to comply with the procedures described in the protocol, including responding to simple questionnaires either by the recipient in person or by a next relative (spouse, parent) who lives with the recipient;
* Patients with good general hygiene;
* Radiographic exam allowing a complete observation of the osseous defect;
* Mimetis approval of the feasibility.

Exclusion Criteria:

* Active tumour;
* Passive tumour with cancer recurrence within 10 years;
* Practice of intensive contact sport exercise during the clinical trial duration;
* Concomitant participation in other clinical trials;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study;
* Women who are breastfeeding;
* Alcohol or drug abuse as noted in subject records or in subject history;
* Patients with a medical condition that may compromise the healing process or history of systemic diseases that would contraindicate the surgical treatment or any other disease that might have an influence on the involved tissues, such as: severe metabolic disorders, osteogenesis imperfecta, osteoporosis, infectious and degenerative bone diseases, immunodeficiency (congenital or acquired), autoimmune disease, Osler-Weber-Rendu syndrome, unbalanced diabetes, transient hypercalcemia, allergic disposition to phosphate calcium components, titanium or collagen etc; immunosuppressive therapy, steroid therapy, heparin treatment, corticoid treatment, treatments that interfere in the calcium-phosphate metabolism, bisphosphonate intake, Paclitaxel treatment, methotrexate medication etc);
* Acute and chronic infections in the surgery area (e.g. soft tissue infections, inflammatory and bacterial osteopathy, osteomyelitis) and / or mucosal diseases in the areas to be treated;
* In case of intraoral surgery, heavy smokers (>10 cigarettes) excluded;
* Inability to return for follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Geometric evolution of the grafted volume through radiological evaluation | 6 months post-surgery

SECONDARY OUTCOMES:
Geometric evolution of the grafted volume through radiological evaluation | 12 months post-surgery
Versatility of MimetikOss 3D patient-specific bone substitute | 12 months post-surgery
  MimetikOss 3D can be implanted to regenerate osseous defect from different indications of the maxillofacial area (dental area, jaw and maxilla reconstruction, zygomatic reconstruction and/or chin reconstruction for instance).
Incidence of serious adverse events and adverse events | during the surgery / 6 months post-surgery / 12 months post-surgery
Bone union observation | 12 months post-surgery
Surgical technique improvement in terms of accuracy of MimetikOss 3D design and positioning | directly after the surgery / 6 months post-surgery / 12 months post-surgery
Surgical technique improvement in terms of total surgery duration and duration of implantation of MimetikOss 3D | during the surgery
Surgical technique improvement in terms of blood loss measurement | during the surgery
Surgical technique improvement in terms of surgeon satisfaction | 12 months post-surgery
Aesthetic evaluation by visual observation of the symmetry of the face, pictures and/or irregular contours prosthetic palpable (if applicable) | directly after the surgery / 6 months post-surgery / 12 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Òscar Escuder i de la Torre, Principal Investigator — University Hospital Parc Taulí Sabadell

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR